CLINICAL TRIAL: NCT01484639
Title: Transfusion Requirements in Cardiac Surgery (TRICS II): A Randomized Controlled Trial
Brief Title: Transfusion Requirements in Cardiac Surgery
Acronym: TRICSII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nadine Shehata (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Health Canada (Other Government)
Responsible Party: Sponsor-Investigator, Nadine Shehata, Principal Investigator-Sponsor, Unity Health Toronto
Organization: Unity Health Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: TRICSII; Application #232416 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2011-11-30; First posted 2011-12-02 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Cardiac Surgery
Keywords: transfusion; cardiac surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Restrictive transfusion triggers (Active Comparator): Patients allocated to a "restrictive" transfusion group will receive a red cell transfusion if their hemoglobin is 75 g/L or less intraoperatively and postoperatively.
  Interventions: Other: Restrictive transfusion triggers
- Liberal transfusion triggers (Active Comparator): Patients allocated to a "liberal" transfusion strategy will receive red cell transfusion if their hemoglobin concentration is 95 g/L or less intraoperatively and postoperatively in the intensive care unit, and less than 85 g/L on the ward.
  Interventions: Other: Liberal transfusion triggers

INTERVENTIONS:
Other: Liberal transfusion triggers — Patients allocated to a "liberal" transfusion strategy will receive red cell transfusion if their hemoglobin concentration is 95 g/L or less intraoperatively and postoperatively in the intensive care unit, and less than 85 g/L on the ward.
  Arms: Liberal transfusion triggers
Other: Restrictive transfusion triggers — Patients allocated to a "restrictive" transfusion group will receive a red cell transfusion if their hemoglobin is 75 g/L or less intraoperatively and postoperatively.
  Arms: Restrictive transfusion triggers

SUMMARY:
This is a multi-centre randomized controlled pilot trial of two transfusion strategies in high risk patients having cardiac surgery. This study will be conducted in 7 Canadian centers and 1 American centre. Patients allocated to a "restrictive" transfusion strategy will receive a red cell transfusion if their hemoglobin is 75 g/L or less intraoperatively and postoperatively. Patients allocated to a "liberal" transfusion strategy will receive red cell transfusion if their hemoglobin concentration is 95 g/L or less intraoperatively and postoperatively in the intensive care unit, and less than 85 g/L on the ward.

The primary objectives of this study are to determine 1) enrollment rates (patients enrolled/patients eligible), 2) consent rates (consent obtained/patients approached); and 3) protocol adherence (incidence and reasons for non adherence, lack of consent, rates of contamination and utilization of co-interventions). The secondary objectives are to determine 1) the mortality rate and the rate of the composite outcome for morbidity of renal, cardiac, neurological and infectious adverse events; 2) the proportion of missing data as a measure of the feasibility of the case report form; and 3) the proportion of blood products utilized (red cells, platelets and plasma).

The results of the multicentre pilot study will be used to 1) maximize enrollment rates to ensure timely completion of recruitment of a definitive large randomized controlled trial, 2) maximize adherence rates, 3) determine event rates for sample size estimation for a definitive study, and to 4) optimize the case report form.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* European System for Cardiac Operative Risk Evaluation (EuroSCORE) of 6 or more
* Consent

Exclusion Criteria:

* Pregnancy
* Refusal of blood products
* Participating in autologous blood donation program
* Based on the preoperative hemoglobin, the predicted hematocrit on cardiopulmonary bypass is greater than 33% (hemoglobin concentration of 110 g/L) or less than 18% (hemoglobin concentration of 60 g/L)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2012-01; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Enrollment rate | baseline
  To determine enrollment rates (patients enrolled/patients eligible), consent rates (consent obtained/patients approached)
Protocol adherence | 28 days or hospital discharge
  To determine protocol adherence (incidence and reasons for non adherence, lack of consent, rates of contamination and utilization of co-interventions).

SECONDARY OUTCOMES:
Mortality and morbidity | 28 days or hospital discharge
  To determine the mortality rate and a composite outcome for morbidity (renal, cardiac, neurological and infectious adverse events).
Missing data | 28 days or hospital discharge
  To determine the proportion of missing data as a measure of the feasibility of the case report form
Blood product utilization | 28 days or hospital discharge
  To determine the proportion of blood products utilized (red cells, platelets and plasma)

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Shehata, MD, Principal Investigator — Li Ka Shing Knowledge Institute, Mount Sinai Hospital; David Mazer, MD, Principal Investigator — Unity Health Toronto
Locations (8):
- Virginia Commonwealth University, Richmond, Virginia, United States
- Canada (7):
  - Foothills Medical Centre, Calgary, Alberta
  - Alberta Health Services, Edmonton, Alberta
  - St. Boniface General Hospital, Winnipeg, Manitoba
  - Hamilton General Hospital, Hamilton, Ontario
  - Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449